CLINICAL TRIAL: NCT06707948
Title: Comparison of Different Treatment Strategies for Root Injury Behind the Medial Meniscus to Delay the Progression of Knee Osteoarthritis: a Prospective Cohort Study
Brief Title: A Study on Different Treatments for Knee Osteoarthritis Caused by Damaged Roots of the Medial Meniscus.
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yinxian Yu, Associate Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: IIT2024-109
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis; Meniscus Lesion
Keywords: posterior meniscus root lesion;Osteoarthrotis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Conservative treatment group: Non-steroidal anti-inflammatory and analgesic drugs
- Arthroscopic partial meniscectomy group: Arthroscopically, the damaged free meniscus is trimmed, ground, and partially resected;
  Interventions: Procedure: Arthroscopic meniscus surgery
- Arthroscopic meniscus suture repair group: Arthroscopic download of the posterior meniscus root injury, placement of sutures through the bone tunnel to fix the meniscus, and then cutting it with a knot to complete the meniscus suture repair.
  Interventions: Procedure: Arthroscopic meniscus surgery

INTERVENTIONS:
Procedure: Arthroscopic meniscus surgery — Comparison of the incidence of osteoarthritis with conservative treatment as well as arthroscopic partial resection as well as arthroscopic repair surgery for a condition known as posterior meniscus root injury.
  Groups: Arthroscopic meniscus suture repair group; Arthroscopic partial meniscectomy group

SUMMARY:
Medial meniscus posterior root tears (MMPRT) account for 20% or more of all meniscus tears, but the diagnosis and treatment of this condition continues to plague the general population due to the complexity of the diagnosis and uncertainty of the treatment. Early as well as timely diagnosis and treatment is one of the effective ways to avoid accelerated knee degeneration. Based on this study, our team is going to conduct a clinical study on posterior medial meniscus tear, combining Magnetic Resonance Imaging(MRI) to dynamically assess the changes of meniscus and articular cartilage surface after the injury, and selecting a specific patient group to carry out different therapeutic interventions, which mainly include conservative treatment, partial meniscectomy, and meniscal repair, in order to clarify the effects of different treatment modalities on the articular cartilage after the posterior meniscus tear, and to help to delay the degeneration of knee joints. This is to clarify the effects of different treatment modalities on the articular cartilage after posterior medial meniscus tears and to provide appropriate advice for delaying the progression of osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of posterior root tear of the medial meniscus;
2. Patients with K-L classification ≤ grade II;
3. The age range of 50-65 years old;
4. International Cartilage Repair Society (ICRS) Modified Magnetic Resonance Imaging Grading System ≤ Grade 2;
5. International Cartilage Repair Society (ICRS) arthroscopic grading system ≤ grade 2;
6. Knee joint mobility ≥90°;
7. Inversion deformity ≤10°;
8. Must be able to complete follow-up MRI within 2 years after knee meniscus surgery;
9. Must be able to complete clinical data;

Exclusion Criteria:

1. Can not participate in this study;
2. Patients with concomitant meniscal injuries elsewhere;
3. knee joint infection disease;
4. Osteoporosis disease;
5. Patients with previous history of knee surgery;
6. Knee joint instability disease;
7. Severe KOA disease;
8. Can not cooperate with MRI detection;
9. Cannot tolerate the surgery;
10. Those who cannot tolerate the arthroscopic knee surgery;
11. Neuromuscular system pathology disease;

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with posterior root injuries of the medial meniscus
Sampling Method: Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
the incidence of KOA | 30th November 2024 -30th November 2027

SECONDARY OUTCOMES:
Articular cartilage T2-mapping value | 30th November 2024 -30th November 2027
  Articular cartilage T2 mapping values, post-standardised range 0-1

OTHER OUTCOMES:
VAS (visual analogue scale)，VAS score | 30th November 2024 -30th November 2027
  The specific scoring method is to draw a 10 cm horizontal line on top of the paper, with 0 at one end of the line indicating no pain, 10 at the other end indicating severe pain, and the middle portion indicating varying degrees of pain.
Lysholm score | 30th November 2024 -30th November 2027
  The score consists of eight indicators: pain (25 points), instability (25 points), atresia (15 points), swelling (10 points), limp (5 points), stair climbing (10 points), squatting posture (5 points), and the use of supports (5 points), with a total score of 100, with higher scores representing better knee function. 95 points or more is considered excellent, 94-85 points is good, 84-65 points is fair, and less than 65 points is poor. A score of less than 65 is poor.
HSS (Hospital for Special Surgery) Score | 30th November 2024 -30th November 2027
  The score is out of 100 and consists of pain (30 points), function (22 points including walking and stair climbing), knee mobility (18 points), muscle strength (10 points), flexion deformity (10 points), joint stability (10 points), and deductions (-5 points). The higher the score, the better the knee function.

IPD SHARING:
Plan to Share IPD: Undecided
Decide whether to share data based on the level of completion of the project

REFERENCES:
- [Background] Jung YH, Choi NH, Oh JS, Victoroff BN. All-inside repair for a root tear of the medial meniscus using a suture anchor. Am J Sports Med. 2012 Jun;40(6):1406-11. doi: 10.1177/0363546512439181. Epub 2012 Mar 16. PMID 22427620
- [Background] Faucett SC, Geisler BP, Chahla J, Krych AJ, Kurzweil PR, Garner AM, Liu S, LaPrade RF, Pietzsch JB. Meniscus Root Repair vs Meniscectomy or Nonoperative Management to Prevent Knee Osteoarthritis After Medial Meniscus Root Tears: Clinical and Economic Effectiveness. Am J Sports Med. 2019 Mar;47(3):762-769. doi: 10.1177/0363546518755754. Epub 2018 Mar 8. PMID 29517925
- [Background] Chung KS, Ha JK, Yeom CH, Ra HJ, Jang HS, Choi SH, Kim JG. Comparison of Clinical and Radiologic Results Between Partial Meniscectomy and Refixation of Medial Meniscus Posterior Root Tears: A Minimum 5-Year Follow-up. Arthroscopy. 2015 Oct;31(10):1941-50. doi: 10.1016/j.arthro.2015.03.035. Epub 2015 Jun 18. PMID 26095821
- [Background] Allaire R, Muriuki M, Gilbertson L, Harner CD. Biomechanical consequences of a tear of the posterior root of the medial meniscus. Similar to total meniscectomy. J Bone Joint Surg Am. 2008 Sep;90(9):1922-31. doi: 10.2106/JBJS.G.00748. PMID 18762653
- [Background] Bin SI, Kim JM, Shin SJ. Radial tears of the posterior horn of the medial meniscus. Arthroscopy. 2004 Apr;20(4):373-8. doi: 10.1016/j.arthro.2004.01.004. PMID 15067276
- [Background] Ozkoc G, Circi E, Gonc U, Irgit K, Pourbagher A, Tandogan RN. Radial tears in the root of the posterior horn of the medial meniscus. Knee Surg Sports Traumatol Arthrosc. 2008 Sep;16(9):849-54. doi: 10.1007/s00167-008-0569-z. Epub 2008 Jun 7. PMID 18536902
- [Background] Nakagawa Y, Mukai S, Sakai S, Nakamura R, Takahashi M, Nakagawa S. Preoperative diagnosis of knee cartilage, meniscal, and ligament injuries by magnetic resonance imaging. J Exp Orthop. 2023 Apr 20;10(1):47. doi: 10.1186/s40634-023-00595-y. PMID 37079120
- [Background] Cao G, Gao S, Xiong B. Application of quantitative T1, T2 and T2* mapping magnetic resonance imaging in cartilage degeneration of the shoulder joint. Sci Rep. 2023 Mar 20;13(1):4558. doi: 10.1038/s41598-023-31644-2. PMID 36941288
- [Background] Ozel MA, Ogul H, Koksal A, Kose M, Tuncer K, Eren S, Kantarci M. Detection of the glenoid bare spot by non-arthrographic MR imaging, conventional MR arthrography, and 3D high-resolution T1-weighted VIBE MR arthrography: comparison with CT arthrography. Eur Radiol. 2023 May;33(5):3276-3285. doi: 10.1007/s00330-023-09443-0. Epub 2023 Feb 16. PMID 36792853
- [Background] Nguyen JC, De Smet AA, Graf BK, Rosas HG. MR imaging-based diagnosis and classification of meniscal tears. Radiographics. 2014 Jul-Aug;34(4):981-99. doi: 10.1148/rg.344125202. PMID 25019436
- [Background] Anz AW, Branch EA, Saliman JD. Biomechanical comparison of arthroscopic repair constructs for meniscal root tears. Am J Sports Med. 2014 Nov;42(11):2699-706. doi: 10.1177/0363546514549445. Epub 2014 Sep 15. PMID 25225682
- [Background] Bhatia S, LaPrade CM, Ellman MB, LaPrade RF. Meniscal root tears: significance, diagnosis, and treatment. Am J Sports Med. 2014 Dec;42(12):3016-30. doi: 10.1177/0363546514524162. Epub 2014 Mar 12. PMID 24623276
- [Background] Lee OS, Lee SH, Lee YS. Comparison of the Radiologic, Arthroscopic, and Clinical Outcomes between Repaired versus Unrepaired Medial Meniscus Posterior Horn Root Tear During Open Wedge High Tibial Osteotomy. J Knee Surg. 2021 Jan;34(1):57-66. doi: 10.1055/s-0039-1692992. Epub 2019 Jul 9. PMID 31288272
- [Background] Krych AJ, Johnson NR, Mohan R, Hevesi M, Stuart MJ, Littrell LA, Collins MS. Arthritis Progression on Serial MRIs Following Diagnosis of Medial Meniscal Posterior Horn Root Tear. J Knee Surg. 2018 Aug;31(7):698-704. doi: 10.1055/s-0037-1607038. Epub 2017 Sep 26. PMID 28950387
- [Background] Hwang BY, Kim SJ, Lee SW, Lee HE, Lee CK, Hunter DJ, Jung KA. Risk factors for medial meniscus posterior root tear. Am J Sports Med. 2012 Jul;40(7):1606-10. doi: 10.1177/0363546512447792. Epub 2012 May 11. PMID 22582224
- [Background] Matheny LM, Ockuly AC, Steadman JR, LaPrade RF. Posterior meniscus root tears: associated pathologies to assist as diagnostic tools. Knee Surg Sports Traumatol Arthrosc. 2015 Oct;23(10):3127-31. doi: 10.1007/s00167-014-3073-7. Epub 2014 May 28. PMID 24866130
- [Background] LaPrade RF, Ho CP, James E, Crespo B, LaPrade CM, Matheny LM. Diagnostic accuracy of 3.0 T magnetic resonance imaging for the detection of meniscus posterior root pathology. Knee Surg Sports Traumatol Arthrosc. 2015 Jan;23(1):152-7. doi: 10.1007/s00167-014-3395-5. Epub 2014 Nov 7. PMID 25377189
- [Background] Bonasia DE, Pellegrino P, D'Amelio A, Cottino U, Rossi R. Meniscal Root Tear Repair: Why, When and How? Orthop Rev (Pavia). 2015 Jun 11;7(2):5792. doi: 10.4081/or.2015.5792. eCollection 2015 Jun 3. PMID 26330993
- [Background] Fujii M, Furumatsu T, Miyazawa S, Kodama Y, Hino T, Kamatsuki Y, Ozaki T. Bony landmark between the attachment of the medial meniscus posterior root and the posterior cruciate ligament: CT and MR imaging assessment. Skeletal Radiol. 2017 Aug;46(8):1041-1045. doi: 10.1007/s00256-017-2625-6. Epub 2017 Mar 18. PMID 28314900
- [Background] Sun D, Neumann J, Joseph GB, Foreman S, Nevitt MC, McCulloch CE, Li X, Link TM. Introduction of an MR-based semi-quantitative score for assessing partial meniscectomy and relation to knee joint degenerative disease: data from the Osteoarthritis Initiative. Eur Radiol. 2019 Jun;29(6):3262-3272. doi: 10.1007/s00330-018-5924-y. Epub 2019 Jan 7. PMID 30617481
- [Background] Marinetti A, Tessarolo F, Ventura L, Falzone A, Neri M, Piccoli F, Rigoni M, Mase M, Cortese F, Nollo G, Della Sala SW. Morphological MRI of knee cartilage: repeatability and reproducibility of damage evaluation and correlation with gross pathology examination. Eur Radiol. 2020 Jun;30(6):3226-3235. doi: 10.1007/s00330-019-06627-5. Epub 2020 Feb 13. PMID 32055948
- [Background] Verma P, Dalal K. Serum cartilage oligomeric matrix protein (COMP) in knee osteoarthritis: a novel diagnostic and prognostic biomarker. J Orthop Res. 2013 Jul;31(7):999-1006. doi: 10.1002/jor.22324. Epub 2013 Feb 19. PMID 23423905
- [Background] Yunus MHM, Nordin A, Kamal H. Pathophysiological Perspective of Osteoarthritis. Medicina (Kaunas). 2020 Nov 16;56(11):614. doi: 10.3390/medicina56110614. PMID 33207632
- [Background] Jacobs JJ, Jevsevar DS, Brown GA, Cummins DS. AAOS Osteoarthritis Guideline: transparency and credibility. Arthroscopy. 2014 Jun;30(6):656-8. doi: 10.1016/j.arthro.2014.03.002. No abstract available. PMID 24862694
- [Background] Su K, Bai Y, Wang J, Zhang H, Liu H, Ma S. Comparison of hyaluronic acid and PRP intra-articular injection with combined intra-articular and intraosseous PRP injections to treat patients with knee osteoarthritis. Clin Rheumatol. 2018 May;37(5):1341-1350. doi: 10.1007/s10067-018-3985-6. Epub 2018 Jan 31. PMID 29388085